CLINICAL TRIAL: NCT00572416
Title: Fatigue in Breast Cancer:A Behavioral Sleep Intervention
Brief Title: Fatigue in Breast Cancer: A Behavioral Sleep Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0140-02-FB; 5R01NR007762-05 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: fatigue; activity-rest; sleep-wake; psychological distress; symptom management
MeSH Terms: conditions — Breast Neoplasms; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Individual Sleep Promotion Plan (Experimental): Four component behavioral sleep intervention comprised of activity-rest, sleep-wake, psychological distress and symptom management. Four components of the Individual Sleep Promotion Plan are: stimulus control, sleep restruction, relaxation, and sleep hygiene.
  Interventions: Behavioral: Individual Sleep Promotion Plan
- 2 Healthy Eating Control (Placebo Comparator): Equal time and attention, information about healthy eating and general conversation
  Interventions: Behavioral: Healthy Eating Control

INTERVENTIONS:
Behavioral: Individual Sleep Promotion Plan — Four components, including activity-rest, sleep-wake, psychological distress, and symptom management. Sleep-wake component has four strategies: stimulus control, sleep restriction, relaxation, and sleep hygiene
  Arms: 1 Individual Sleep Promotion Plan
Behavioral: Healthy Eating Control — Equal time and attention and information about healthy eating
  Arms: 2 Healthy Eating Control

SUMMARY:
1. This randomized clinical trial compares a four component behavioral sleep intervention group to an attention control healthy eating group
2. The behavioral sleep intervention is designed to reduce fatigue in women with stages I-IIIA breast cancer receiving anthracycline-based chemotherapy
3. The intervention uses an Individual Sleep Promotion Plan to promote daytime activity and nighttime sleep,and to decrease physchological and symptom distress
4. The healthy eating group receives equal time and attention and information on healthy eating
5. All participants receive a research nurse visit 2 days prior to each chemotherapy treatment, and 30, 60, 90 days after the last treatment, and one-year after the first treatment.
6. Adherence to the intervention is calculated at each time
7. Reliable and valid instruments are used, including wrist actigraphy

DETAILED DESCRIPTION:
Higher fatigue levels are found in women with stage I, II or IIIA breast cancer receiving adjuvant chemotherapy (CT) who adopt patterns of daytime inactivity and nighttime restlessness and have more symptom and psychological distress. Interventions that improve sleep quality and reduce daytime fatigue in persons with insomnia may also benefit women receiving adjuvant CT. Using selected factors from Piper's Integrated Fatigue Model (IFM), a randomized, controlled clinical trial will compare women with breast cancer who receive a four component behavioral sleep intervention to women in the attentional control group during and after adjuvant CT. The intervention is designed to reduce fatigue in these women by promoting daytime activity, improving sleep quality and decreasing symptom and psychological distress. The aims of this study are to: 1) Compare the immediate (sleep/wake, activity/exercise, symptoms, psychological distress) and consequent (fatigue) outcomes of women who receive a four component behavioral sleep intervention (sleep hygiene counseling, relaxation therapy, sleep restriction and stimulus control) (n=110) with the outcomes in the healthy eating group (n=110) in women with stage I, II or IIIA breast cancer during 4 or 8 cycles of adjuvant chemotherapy, at 30, 60 and 90 days after their last treatment, and 1 year after their first treatment; 2) Determine the extent to which factors selected from the IFM influence fatigue intensity levels a) in the total sample at baseline and b) differentially influence fatigue intensity levels between groups 30 days after the last chemotherapy treatment and 1 year after the first treatment and 3) Evaluate the adherence to the refined behavioral sleep intervention and preferences for sleep hygiene and relaxation therapy techniques in the experimental group over time. Women will be randomized on the basis of good or poor sleeping history and intent to treat (4 versus 8 cycles of CT) to the intervention or attentional control group. Using the co-scientist model, the sleep intervention group will follow an Individual Sleep Promotion Plan negotiated with the investigator with regularly scheduled reinforcements and revisions. The healthy eating group will receive equal time and attention regarding general topics and nutrition. Established instruments include the Piper Fatigue Scale, Hospital Anxiety and Depression Scale, SF-36 Health Survey, Symptom Experience Scale, Daily Diary and Pittsburgh Sleep Quality Index. Objective measures include wrist actigraph, hemoglobin/ hematocrit, white blood count, T4 & TSH, and body mass index and a C - reactive protein at 1 year. Statistical analyses include RM-ANOVA, generalized estimation equation methodology and multiple regression analysis. Results may inform development of clinical guidelines for fatigue management during adjuvant CT.

ELIGIBILITY:
Inclusion Criteria:

* Ages 19 and older
* Diagnosed for the first time with stage I-IIIA breast cancer
* Post-operative for breast cancer
* Scheduled to receive anthracycline-based adjuvant chemotherapy with our without taxane chemotherapy
* English speaking
* Karnofsky performance Scale score equal to or greater than 60

Exclusion Criteria:

* Comorbid diagnosis of chronic insomnia
* Sleep apnea or chronic fatigue syndrome
* Unstable congestive heart failure
* Chronic obstructive pulmonary disease
* Insulin-depenent diabetes
* Neruomuscular disease
* Abnormal thryoid function
* Depression, or
* Treatment with steriods
* Erratic sleep schedule due to working rotating shifts

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2003-04-01 (Actual); Study Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
Fatigue | 1 year
  Fatigue as measured by Piper Fatigue Scale

SECONDARY OUTCOMES:
Activity-rest as measured by SF-36v2 and actigraphy | 1 year
  Activity-rest as measured by SF-36v2 and actigraphy
Sleep-wake | 1 year
  Sleep-wake as measured by Pittsburgh Sleep Quality Index and actigraphy
Psychological mood | 1 year
  Psychological mood as measured by Hospital Anxiety and Depression Scale
Symptom experience | 1 year
  Symptom experience as measured by Symptom Experience Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Berger, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Berger AM, Farr LA, Kuhn BR, Fischer P, Agrawal S. Values of sleep/wake, activity/rest, circadian rhythms, and fatigue prior to adjuvant breast cancer chemotherapy. J Pain Symptom Manage. 2007 Apr;33(4):398-409. doi: 10.1016/j.jpainsymman.2006.09.022. PMID 17397701
- [Result] Berger AM, Neumark DE, Chamberlain J. Enhancing recruitment and retention in randomized clinical trials of cancer symptom management. Oncol Nurs Forum. 2007 Mar;34(2):E17-22. doi: 10.1188/07.ONF.E17-E22. PMID 17573292